CLINICAL TRIAL: NCT00418925
Title: Phase II, Double Blind, Randomized, Placebo Controlled Trial of Dronabinol for the Treatment of Cervical Dystonia
Brief Title: Efficacy of Dronabinol for the Treatment of Cervical Dystonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Dystonia Medical Research Foundation (Other)
Responsible Party: Susan Fox, UHN Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MDC DRO 2006
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2007-08

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dronabinol — 2.5 mg tablets; titrated over 14 days and 7 days steady dose
  Other Names: Marinol(R)

SUMMARY:
Cervical dystonia (CD) is characterized by abnormal, involuntary sustained cervical muscles contractions associated with twisting movements and abnormal postures of the neck that can be quite disabling. Currently there are no good oral medications for the treatment of CD. While botulinum toxin injections are effective in most, they require repeat injections and there are some patients who either stop responding or who never respond at all. Therefore, better treatments are needed. While the underlying mechanisms of dystonia are not entirely known, there is some information suggesting that it is ude to an underactivity of a chemical compound, GABA, that is located in the basal ganglia. Cannabinoids are a compound than can enhance transmission of GABA, and thus, may alleviate the symptoms of dystonia. Dronabinol, one such cannabinoid, has been widely used to treat anorexia and nausea in chemotherapeutic patients. The aim of this study, therefore, is to study the effect of dronabinol on cervical dystonia

DETAILED DESCRIPTION:
The study is a double-blind, randomized, placebo-controlled, crossover, phase II study of dronabinol versus placebo. Thirty patients with idiopathic cervical dystonia will be enrolled in the study. Patients will be randomized to either dronabinol or placebo by a computer-generated random numbers table that will be kept in the central pharmacy until the end of the trial. Only the central pharmacy will be aware of treatment allocation; all others will be blinded for the duration of the trial.

Regardless of treatment allocation, study participants will begin taking their assigned study medications on Day 1, increasing the "dose" (actual increase in dose for dronabinol-assigned arm, fictional increase in dose for placebo-assigned arm) every 3 days. At the end of the third week, on Day 21, the study participant will complete the first phase of study medication and remain off study medication for a period of two weeks, and will have a planned study visit. On Day 36, the study participant will have a planned study visit, the new medication will be dispensed, and the participant will begin taking the other arm of the study medication for a period of 3 weeks, in the same manner as the first arm. At the end of the 3 weeks (8 weeks in total), the study participant will discontinue the assigned study medication and will attend a planned study visit for study termination. At each visit, patients will be assessed with a medical and neurological history and examination and a video recording made for post hoc analysis of TWSTRS by a rater blinded to the treatment arm.

The main issue with compliance to study medication will relate to side-effects. Side-effects are mainly dose related and can be minimized with a dose escalation protocol, which is planned in this study. Compliance and adverse effects will be monitored by weekly phone calls for side effects and pill counts at the end of each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year old male and female patients with idiopathic cervical dystonia -

Exclusion Criteria:

* Secondary causes of dystonia; history of substance abuse, psychosis, ischemic heart disease, symptomatic postural hypotension, liver disease (LFTs > 2 times normal), renal disease
* Women who are pregnant or plan on becoming pregnant during the course of the trial
* Use of botulinum toxin as a treatment for cervical dystonia in the preceding 4 months
* Use of other GABA mediated drugs including: gabapentin, phenobarbital, benzodiazepines, or baclofen
* Use of other cannabinoids in the preceding month
* Refusal to refrain from use of other cannabinoid compounds during the course of the trial
* Refusal to refrain from operating heavy machinery or driving during the course of the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)with 3 weeks of active treatment compared to placebo | beginning and end of each treatment

SECONDARY OUTCOMES:
To determine the rate and severity of adverse events within and between participants | Beginning and end of each treatment
To observe changes within and between participants in the Global Impression Scale (GIS) | End of each treatment
To observe changes within and between participants in the Visual Analog Pain Scale | beginning and end of each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Fox, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada